CLINICAL TRIAL: NCT02992691
Title: Dose Response of Three Experimental Dentifrices in Plaque Removal in a Single Brushing Model
Brief Title: Efficacy of Three Experimental Toothpastes to Remove Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206886
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

ARMS (5):
- Test Product 1 (Experimental): Participants will be instructed to dose a toothbrush with full ribbon of dentifrice. Participants will brush their teeth once for one timed minute.
  Interventions: Drug: 20% w/w sodium bicarbonate
- Test Product 2 (Experimental): Participants will be instructed to dose a toothbrush with full ribbon of dentifrice. Participants will brush their teeth once for one timed minute.
  Interventions: Drug: 35% w/w sodium bicarbonate
- Test Product 3 (Experimental): Participants will be instructed to dose a toothbrush with full ribbon of dentifrice. Participants will brush their teeth once for one timed minute.
  Interventions: Drug: 50% w/w sodium bicarbonate
- Positive Control (Active Comparator): Participants will be instructed to dose a toothbrush with full ribbon of dentifrice. Participants will brush their teeth once for one timed minute.
  Interventions: Drug: 67% w/w sodium bicarbonate
- Negative Control (Other): Participants will be instructed to dose a toothbrush with full ribbon of dentifrice. Participants will brush their teeth once for one timed minute.
  Interventions: Drug: 0% w/w sodium bicarbonate

INTERVENTIONS:
Drug: 20% w/w sodium bicarbonate — Dentifrice containing 20% w/w sodium bicarbonate.
  Arms: Test Product 1
Drug: 35% w/w sodium bicarbonate — Dentifrice containing 35% w/w sodium bicarbonate.
  Arms: Test Product 2
Drug: 50% w/w sodium bicarbonate — Dentifrice containing 20% w/w sodium bicarbonate.
  Arms: Test Product 3
Drug: 67% w/w sodium bicarbonate — Dentifrice containing 67% w/w sodium bicarbonate.
  Arms: Positive Control
Drug: 0% w/w sodium bicarbonate — Dentifrice containing 0% sodium bicarbonate and 1450 parts per million (ppm) fluoride.
  Arms: Negative Control

SUMMARY:
The Dose response of three experimental toothpastes (test product 1, test product 2 and test product 3) to remove plaque after a single brushing, compared to a positive control and negative control dentifrice will be evaluated.

DETAILED DESCRIPTION:
This will be a single centre, controlled, examiner blind, five treatment, five period, crossover design study in healthy participants. This study will evaluate the dose response of three experimental toothpastes (test product 1, test product 2 and test product 3) to remove plaque after a single brushing, compared to a positive control and negative control dentifrice. Plaque removal efficacy will be measured by Turesky modification of Quigley Hein Plaque Index (TPI).

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18- 65 years
* Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or oral/dental examination. Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Good dental health based on medical history and oral soft tissue examination at screening, a minimum of 20 permanent gradable teeth (Gradable teeth are those where restorative materials cover less than 25% of the tooth surface to be graded), and mean Turesky plaque score of ≥ 2.00 at Visit 1 and Visit 2 (pre-brushing plaque assessment).
* Understands and is willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study: cosmetic studies within 14 days of the screening visit or receipt of an investigational drug within 30 days of the screening visit and previous participation in this study.
* Recent history (within the last year) of alcohol or other substance abuse.
* An employee of the sponsor or the study site or members of their immediate family and an employee of any toothpaste manufacturer or their immediate family.
* Antibiotic treatment within 14 days prior to Visit 2 or throughout the study, any other treatment that would interfere with the study outcomes, at the discretion of the examiner or investigator.
* High levels of extrinsic stain or calculus deposits which might interfere with plaque assessments at the discretion of the investigator, dental conditions / disease requiring immediate treatment, pre-existing sensitivity to oral care products, severe gingivitis that may, in the opinion of the investigator, compromise the study or the oral health of the participants if they participate in the study, presence of orthodontic bands or appliances, extensive crowns, partial dentures, or fixed retainers on the maxillary or mandibular teeth, active carious lesions needing immediate care, oral lesions/manifestations that would impact on the outcome of the study, presence of oral or peri-oral ulceration including herpetic lesions at the time of screening, have current active caries or periodontitis that may, in the opinion of the investigator, compromise the study or the oral health of the participants if they participate in the study, restorations in a poor state of repair that may, in the opinion of the investigator, compromise the study or the oral health of the participants if they participate in the study, use of a chlorhexidine mouthwash within 14 days of Visit 2 or through the study and current use of Listerine, Corsodyl or any antimicrobial mouth rinse or throughout the study.
* Participant unwilling to abstain from using chewing tobacco (with or without tobacco) and Participant unwilling to abstain from smoking tobacco or E-cigarettes for 4 hours prior to all visits and until all dental assessments are completed at each visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

REFERENCES:
- [Result] Jose A, Parkinson CR, Manger C, Bielfeldt S, Krause C. Randomized Clinical Dose-Response Study to Evaluate Plaque Removal by Three Experimental Sodium Bicarbonate Toothpastes Using a Single Brushing Model. J Clin Dent. 2018 Dec;29(4):75-80. PMID 30942962
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206886&attachmentIdentifier=b79c83c9-8d09-4165-888d-5b5838a48e61&fileName=gsk-206886-clinical-study-report-redact.pdf&versionIdentifier=
- See also: Randomized Clinical Dose-Response Study to Evaluate Plaque Removal by Three Experimental Sodium Bicarbonate Toothpastes Using a Single Brushing Model. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Dose+Response+of+Three+Experimental+Dentifrices+in+Plaque+Removal+in+a+Single+Brushing+Model

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in Germany
Pre-assignment Details: A total of 100 participants were screened, out of which 25 participants were screening failure. Remaining 75 participants were enrolled in the study. Out of 75 enrolled participants, 6 did not meet eligibility criteria, 3 withdrew their consent, 10 participants, due to other reason (not specified). Remaining 56 were randomized in the study.
Groups:
- Overall Study: This was a single-center, controlled, examiner-blind, five-treatment, five-period, crossover design study in healthy volunteers. Each participant received Test Product 1 (Dentifrice containing 20 percent [%] weight by weight [w/w] sodium bicarbonate), Test product 2 (Dentifrice containing 35% w/w sodium bicarbonate) Test product 3 (Dentifrice containing 50% w/w sodium bicarbonate), positive control (Dentifrice containing 67% w/w sodium bicarbonate) and negative control (Dentifrice containing 0% sodium bicarbonate and 1450 parts per million (ppm) fluoride).
Period: Overall Study
Arm/Group | Overall Study
Started | 56
Received Test Product 1 | 55
Received Test Product 2 | 55
Received Test Product 3 | 52
Received Positive Control | 55
Received Negative Control | 55
Completed | 53
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This was five-treatment, five-period, crossover design study. Each participant received Test Product 1 (Dentifrice containing 20 percent [%] weight by weight [w/w] sodium bicarbonate), Test product 2 (Dentifrice containing 35% w/w sodium bicarbonate) Test product 3 (Dentifrice containing 50% w/w sodium bicarbonate), positive control (Dentifrice containing 67% w/w sodium bicarbonate) and negative control (Dentifrice containing 0% sodium bicarbonate and 1450 parts per million [ppm] fluoride).
Arm/Group | Overall Study
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.3 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Pre-brushing) After a Single Brushing Treatment (Post-brushing) Turesky Modification of Quigley Hein Plaque Index (TPI), Positive Control Versus [vs.] Negative Control
Description: The dental examiner used Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth.Overall plaque scores were calculated taking average over all tooth sites for participant.Plaque was first disclosed using dye solution followed by disclosing solution.They expectorated and rinsed with 10 milliliters (mL) water for 10 seconds (sec),expectorated again. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial,facial,distofacial,mesiolingual,lingual,distolingual surfaces.Disclosed plaque was scored for each tooth surface separately as:0 No plaque;1 Slight flecks of plaque at cervical margin of the tooth;2 A thin continuous band of plaque(1 mm or smaller) at cervical margin of tooth;3 A band of plaque wider than 1 mm but covering less than 1/3 of the crown of tooth;4 Plaque covering at least 1/3 but less than 2/3 of crown of tooth;5 Plaque covering 2/3 or more of crown of tooth. Score range 0-5.Lower scores indicate less plaque area.
Time Frame: Up to 5 weeks
Population: Intent to treat (ITT) population was the primary population of analysis. The ITT population was defined as those participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Positive Control: Participant applied a full ribbon of dentifrice containing 67% w/w sodium bicarbonate and brushed their teeth for one timed minute.
- Negative Control: Participant applied a full ribbon of dentifrice containing 0% sodium bicarbonate and 1450 ppm fluoride and brushed their teeth for one timed minute.
Arm/Group | Positive Control | Negative Control
Number analyzed (Participants) | 55 | 55
Score on a Scale | -0.57 (0.247) | -0.54 (0.253)
Statistical Analysis 1: Comparison: Positive Control vs Negative Control; This comparison was tested under a null hypothesis of no difference against alternative hypothesis of a difference between treatments; Test type: Other; p = 0.6674, ANCOVA — From ANCOVA analysis for change from pre-brushing with treatment and period as fixed effect, participant as random effect, participant-level baseline and period level minus participant-level baseline as covariates; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.06 to 0.04]

2. Secondary Outcome: Change From Baseline (Pre-brushing) After a Single Brushing Treatment (Post-brushing) Turesky Modification of Quigley Hein Plaque Index (Test Product 1, 2 and 3 vs Negative Control)
Description: The dental examiner used Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth.Overall plaque scores were calculated taking average over all tooth sites for participant.Plaque was first disclosed using dye solution followed by disclosing solution.They expectorated and rinsed with 10 mL of water for 10 sec,expectorated again. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial,facial,distofacial,mesiolingual,lingual,distolingual surfaces.Disclosed plaque was scored for each tooth surface separately as:0 No plaque;1 Slight flecks of plaque at cervical margin of the tooth;2 A thin continuous band of plaque(1 mm or smaller) at cervical margin of tooth;3 A band of plaque wider than 1 mm but covering less than 1/3 of the crown of tooth;4 Plaque covering at least 1/3 but less than 2/3 of crown of tooth;5 Plaque covering 2/3 or more of crown of tooth. Score range 0-5.Lower scores indicate less plaque area.
Time Frame: Up to 5 weeks
Population: ITT population was the primary population of analysis. The ITT population was defined as those participants who were randomized, received at least one dose of study product and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Test Product 1: Participant applied a full ribbon of dentifrice containing 20% w/w sodium bicarbonate and brushed their teeth for one timed minute.
- Test Product 2: Participant applied a full ribbon of dentifrice containing 35% w/w sodium bicarbonate and brushed their teeth for one timed minute.
- Test Product 3: Participant applied a full ribbon of dentifrice containing 50% w/w sodium bicarbonate and brushed their teeth for one timed minute.
- Negative Control: Participant applied a full ribbon of dentifrice containing 0% w/w sodium bicarbonate and 1450 ppm fluoride brushed their teeth for one timed minute.
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Negative Control
Number analyzed (Participants) | 55 | 52 | 55 | 55
Score on a scale | -0.56 (0.250) | -0.55 (0.231) | -0.55 (0.243) | -0.54 (0.253)

3. Secondary Outcome: Change From Baseline (Pre-brushing) After a Single Brushing Treatment (Post-brushing) Turesky Modification of Quigley Hein Plaque Index (Test Product 1, 2 and 3 vs Positive Control)
Description: The dental examiner used Turesky Modification of the Quigley Hein Index to assess plaque on all gradable teeth.Overall plaque scores were calculated taking average over all tooth sites for participant.Plaque was first disclosed using dye solution followed by disclosing solution.They expectorated and rinsed with 10 mL of water for 10 sec,expectorated again. Plaque was assessed with each tooth being divided into 6 areas including mesiofacial,facial,distofacial,mesiolingual,lingual,distolingual surfaces.Disclosed plaque was scored for each tooth surface separately as:0 No plaque;1 Slight flecks of plaque at cervical margin of the tooth;2 A thin continuous band of plaque(1 mm or smaller) at cervical margin of tooth;3 A band of plaque wider than 1 mm but covering less than 1/3 of the crown of tooth;4 Plaque covering at least 1/3 but less than 2/3 of crown of tooth;5 Plaque covering 2/3 or more of crown of tooth.Score range 0-5.Lower scores indicate less plaque area.
Time Frame: Up to 5 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Positive Control
Number analyzed (Participants) | 55 | 55 | 52 | 55
Score on a scale | -0.56 (0.250) | -0.55 (0.231) | -0.55 (0.243) | -0.57 (0.247)

ADVERSE EVENTS:
Time Frame: Up to 5 weeks
Arm/Group | Test Product 1 | Test Product 2 | Test Product 3 | Positive Control | Negative Control
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/52 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 5/55 | 2/55 | 8/52 | 6/55 | 6/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/52 | 0/55 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product 1 (N=55) | Test Product 2 (N=55) | Test Product 3 (N=52) | Positive Control (N=55) | Negative Control (N=55)
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 2 | 1 | 1
Oral Herpes (Infections and infestations) | 1 | 0 | 2 | 2 | 2
Angular Cheilitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pulpitis Dental (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gingival Erythema (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 1
Oral Mucosal Erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Tongue Coated (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Tonsillar Erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT02992691/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT02992691/SAP_001.pdf